CLINICAL TRIAL: NCT00573092
Title: Genome-Wide Case-Only Study of Antihypertensive Drug-Gene Interactions
Brief Title: Analyzing Gene Regions That May Interact With the Effectiveness of High Blood Pressure Drugs
Status: Withdrawn | Type: Observational
Why Stopped: Withdrawn
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Bruce Psaty, Professor, Medicine & Epidemiology, University of Washington
Other Study IDs: 1411; R01HL085251-01A1 (NIH)
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Myocardial Infarction; Cerebrovascular Accident; Death, Sudden, Cardiac
Keywords: Cardiovascular Epidemiology; Genomics; Genome-Wide Association Study
MeSH Terms: conditions — Myocardial Infarction; Stroke; Death, Sudden, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Data and specimens from three large population-based studies of heart attack, sudden death, and stroke in people treated for high blood pressure with one of the four major classes of high blood pressure drugs

SUMMARY:
High blood pressure is one of the most common health problems in the United States. There are many drug treatment options for high blood pressure, but these medications are not always effective. People with treated high blood pressure can still suffer from other serious cardiovascular health problems, including heart attack, sudden death, or stroke. Genetic variations may cause some people to be more susceptible to these cardiovascular outcomes despite treatment. This study will identify new gene regions that may influence the effectiveness of high blood pressure drugs in preventing the above mentioned cardiovascular conditions.

DETAILED DESCRIPTION:
High blood pressure affects nearly one in three individuals in the United States. There are many factors that can cause high blood pressure, including family history and genetic traits, kidney disease, stress, diabetes, and diet. If left untreated, high blood pressure can increase one's risk for stroke, heart attack, and heart failure. There are four major classes of drugs used to treat high blood pressure, which include diuretics, beta blockers, angiotensin converting enzyme (ACE) inhibitors, and calcium antagonists. Each class works differently in treating high blood pressure, and certain gene regions may affect the effectiveness of the various high blood pressure drugs. The purpose of this study is to identify new gene regions that may influence the effectiveness of the four major high blood pressure drug types in preventing a heart attack, sudden death, or stroke.

This study will draw upon specimens and data from three large population-based studies: the Group Health population, the Cardiovascular Heart Study, and the Jackson Heart Study. New samples of DNA and laboratory data will only be collected from participants in the Group Health population. The remaining samples will be pre-existing samples from the other two studies. Through a whole-genome study of the DNA samples, researchers will distinguish genomic regions of interest for the four major drug classes to identify associations between the drugs and genes in the population. Researchers will further genotype the "interesting" genomic regions discovered in the whole-genome study. Ethnic-specific genetic variations will also be identified to fully characterize the genetic variations. The study will be replicated to assess the validity of the findings.

ELIGIBILITY:
Inclusion Criteria:

* Experience of a first heart attack, stroke, or sudden death
* Member of the Group Health Center (GHC) treated for high blood pressure
* Enrolled at least 1 year in one of the three study populations
* Treated for high blood pressure with one of the four major classes of high blood pressure drugs (diuretics, beta-blockers, ACE inhibitors, or calcium antagonists)

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data and specimens for this study will be collected from three population-based studies: Group Health population, Cardiovascular Heart Study, and Jackson Heart Study. The Group Health population will provide new DNA samples; the Cardiovascular Heart and Jackson Heart studies will provide existing DNA specimens to replicate the study findings from the Group Health population. The Cardiovascular Heart Study involves Americans over the age of 65. The Jackson Heart Study is a cardiovascular disease study in African Americans.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Genomic regions for each of the four major drug classes that influence drug and gene interaction | Measured at completion of genetic analysis

SECONDARY OUTCOMES:
Ethnic-specific genetic variations for each of the four major drug classes that influence drug and gene interaction | Measured at completion of genetic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Bruce M. Psaty, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- Cardiovascular Health Research Unit, Seattle, Washington, United States